CLINICAL TRIAL: NCT03861442
Title: Front-End Processing 3.0 - Noise Reduction, Transient Reduction, Scene Classifier
Brief Title: Front-End Processing 3.0
Acronym: FEP3
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EL_CRD_2017_06
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: front-end features; speech perception; patient reported outcome; Cochlear implants; post lingual sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Adult unilateral MED-EL Cochlear implant users (≥ 6 months), with post-lingual, severe to profound sensory-neural hearing loss.
  Interventions: Device: Audio processor SONNET; Device: SONNET 2: Configuration 1; Device: SONNET 2: Configuration 2; Device: SONNET 2: Configuration 3; Device: SONNET 2: Configuration 4; Device: SONNET 2: OPUS 2 configuration; Device: SONNET 2: SONNET configuration

INTERVENTIONS:
Device: Audio processor SONNET — AI - N/A, WNR - Mild, Beam-former - NAT, AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - N/A, TNR - N/A
  Other Names: Default
Device: SONNET 2: Configuration 1 — AI - Off, WNR - Mild, Beam-former - NAT, AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - Mild, TNR - Mild
Device: SONNET 2: Configuration 2 — AI - Off, WNR - Mild, Beam-former - NAT, AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - Strong, TNR - Strong
Device: SONNET 2: Configuration 3 — AI - Mild, WNR - Mild, Beam-former - Auto (NAT), AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - Auto (Off-Mild), TNR - Auto (Off-Mild)
Device: SONNET 2: Configuration 4 — AI - Strong, WNR - Strong, Beam-former - Auto (OMNI-ABF), AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - Auto (Off-Strong), TNR - Auto (Off-Strong)
Device: SONNET 2: OPUS 2 configuration — AI - Off, WNR - Off, Beam-former - OMNI, AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - N/A, TNR - N/A
Device: SONNET 2: SONNET configuration — AI - Off, WNR - Mild, Beam-former - NAT, AGC Compression - 3:1, AGC Sensitivity - 75%, ANR - N/A, TNR - N/A

SUMMARY:
This study investigated the impact of Automatic Sound Management 3.0 (i.e. ambient noise reduction, transient noise reduction and an adaptive intelligence) as implemented in the SONNET2 on CI users' speech performance and their subjective quality of hearing and device handling.

DETAILED DESCRIPTION:
MED-EL Cochlear Implants (CI) provide auditory sensations via electrical stimulation of the auditory pathways for severely to profoundly hearing-impaired individuals who obtain little or no benefit from acoustic amplification in the best aided condition. Front-end processing of acoustic signals picked up by the audio processor is routinely applied to provide optimal hearing performance under varying listening conditions. Automatic Sound Management (ASM) was introduced by MED-EL with the TEMPO+ audio processor and provided advanced compression and automatic gain management. With the SONNET audio processor, MED-EL introduced ASM 2.0, which added wind noise reduction and microphone directionality to the front-end processing. With the new SONNET2 audio processor, ASM 3.0 was implemented and the features ambient noise reduction, transient noise reduction and an adaptive intelligence (AI) were added.

This study investigated the impact of ASM 3.0 as implemented in the SONNET2 on CI users' speech performance and their subjective quality of hearing.

Subjects' speech performance was tested in quiet (Freiburg Monosyllables Test) and noise (OLSA) with the SONNET audio processor and the SONNNET 2 audio processor (OPUS 2 Configuration, SONNET Configuration, SONNET 2 Configurations 1-4). Additionally, quality of hearing with two questionnaires (HISQUI19, SSQ12) was evaluated with the subjects SONNET and the SONNET 2 configurations 1-4. Device handling with the SONNET and the SONNET 2 audio processor was investigated with a questionnaire (APSQ). Additionally, the data logging function of the SONNET2 audio processor was used to investigate differences in the use of the SONNET configuration and the SONNET 2 configurations 1-4. Subjects were asked to rate the SONNET 2 configurations 1-4 against the SONNET configuration with a product-specific SONNET2 questionnaires. Further, subjective sound quality was evaluated in different auditory settings and subjects' subjective listening effort was evaluated using the ACAES test with the SONNET 2 (OPUS configuration, SONNET configuration, SONNET 2 configuration 1&2).

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 18 years old
* Experienced user (≥ 6 months) of a MED-EL cochlear implant (CI; C40+ and later model)
* Experienced user of a MED-EL SONNET audio processor (≥ 6 months)
* Post-lingual onset of bilateral severe to profound sensory-neural hearing loss
* Unilateral CI user
* A minimum of 10 active electrodes
* A minimum of 40% speech recognition in the Freiburg Monosyllables test in quiet at 65 dB sound pressure level (SPL; at the last time tested)
* Fluent in German (the language of the test centre)
* Signed and dated Informed Consent Form before the start of any study-specific procedure.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* CI user with contralateral hearing equal to or better than 60 dB (PTA measured at 500, 1000, and 2000Hz)
* User with electric-acoustic stimulation (EAS; user of an EAS audio processor)
* Implanted with C40X and C40C
* Implanted with an Auditory Brainstem Implant or Split electrode array
* Known allergic reactions to components of the investigational medical device
* Unstable psychological status
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-lingually deafened adult cochlear implant users with a MED-EL device
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Speech in noise | 8 weeks
  Oldenburg Sentence Test in noise (S0N0)

SECONDARY OUTCOMES:
Speech in quiet | 8 weeks
  Freiburg Monosyllabic test in quiet
Speech in noise | 8 weeks
  Oldenburg Sentence Test in noise (S0N0)
Speech in noise | 8 weeks
  Oldenburg Sentence Test in noise (S0N0T0)
Speech in noise | 8 weeks
  Oldenburg Sentence Test in noise (S0, ±N45, ± N135)
Quality of hearing | 8 weeks
  Hearing Implant Sound Quality Index
Quality of hearing | 8 weeks
  Questionnaire: The Speech, Spatial and Qualities of Hearing Scale (SSQ12; short version, 12 items) with a scale range 0 (worst) to 10 (best)
Device handling | 8 weeks
  Audio Processor Satisfaction Questionnaire (APSQ) with a scale range 0 (worst) to 10 (best)
Subjective Ratings | 8 weeks
  Adaptive CAtegorical Listening Effort Scaling (ACALES); Subjectively perceived listening Effort is evaluated using a 14-step scale contains eight labelled categories (from "effortless" to "extremely strenuous" and "noise only")
Subjective Ratings | 8 weeks
  Subjective Sound Quality Rating
User Satisfaction | 8 weeks
  A product specific questionnaire will be used to gain user satisfaction on the new audio processor and individual setting preferences
Device Use | 8 weeks
  Data Logging
Sound Quality and Quality of hearing | 8 weeks
  Hearing Implant Sound Quality Index 19 (HISQUI19) with a 7-point rating scale (never to always)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Hals-, Nasen- und Ohrenkrankheiten, plastische und ästhetische Operationen, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurz A, Rak K, Hagen R. Improved performance with automatic sound management 3 in the MED-EL SONNET 2 cochlear implant audio processor. PLoS One. 2022 Sep 15;17(9):e0274446. doi: 10.1371/journal.pone.0274446. eCollection 2022. PMID 36108069
- See also: Results of the study, published in an article — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0274446

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03861442/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03861442/SAP_001.pdf